CLINICAL TRIAL: NCT01666405
Title: A Prospective, Multicenter Trial to Investigate the Safety and Efficacy of Percutaneous Tibial Nerve Stimulation for the Treatment of Fecal Incontinence
Brief Title: Prospective, Multicenter Trial to Investigate the Safety and Efficacy of Percutaneous Tibial Nerve Stimulation for the Treatment of Fecal Incontinence
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: business reasons
Sponsor: Uroplasty, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPC032012
Record Dates: First submitted 2012-08-10; First posted 2012-08-16 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Fecal Incontinence
Keywords: Fecal Incontinence; Bowel Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Urgent(R) PC Neuromodulation System (Experimental): Urgent(R) PC Neuromodulation System
  Interventions: Device: Urgent(R) PC Neuromodulation System

INTERVENTIONS:
Device: Urgent(R) PC Neuromodulation System — The Urgent PC Neuromodulation System (Uroplasty, Inc., Minnetonka, MN, USA), device, is an easily administered neuromodulation system designed to deliver retrograde access to the sacral nerve through percutaneous electrical stimulation of the tibial nerve. This method of treatment is referred to as percutaneous tibial nerve stimulation (PTNS).

SUMMARY:
The purpose of this study is to determine the effectiveness of percutaneous tibial nerve stimulation (PTNS) therapy with the Urgent® PC Neuromodulation System (Uroplasty, Inc., Minnetonka, MN, USA) for the treatment of fecal incontinence (FI).

DETAILED DESCRIPTION:
Pilot Study

ELIGIBILITY:
Inclusion Criteria:

* Patient history of chronic FI of more than staining for at least 6 months; staining defined as less than the size of a 25¢ piece (quarter)
* Patient reported and/or failed ≥ 2 conservative therapies (e.g., diet/fiber modification, anti-diarrheal medication, pelvic floor muscle training, biofeedback, medical management, etc.)

Exclusion Criteria:

* Pregnancy or intention to become pregnant during the course of the study
* Implanted electro-medical device (i.e., pacemaker, defibrillator, deep brain stimulator, etc.)
* Clinically significant neurological diseases or nerve damage impacting tibial nerve or pelvic floor function
* Prone to excessive bleeding or bleeding diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness | 18 weeks
  To assess the effectiveness of PTNS by measuring the proportion of patients with ≥50% decrease in the number of fecal incontinence episodes per week based on the results of the 14-day bowel diary at 18 weeks compared to baseline
Safety | 18 weeks
  To characterize adverse events experienced throughout the study

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - UCSF Center for Colorectal Surgery, San Francisco, California
  - Minnesota Colon and Rectal Surgery Associates, Ltd., Minneapolis, Minnesota
  - The Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - Colorectal Surgical Asociates, Houston, Texas
  - Providence Health and Services, Spokane, Washington